CLINICAL TRIAL: NCT04507230
Title: Assessment of COVID-19 Associated Coagulopathy and Hypercoagulable State in Upper Egypt
Brief Title: COVID-19 Associated Coagulopathy in Egypt
Status: Completed | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Azza Abdelaal, lecturer of clinical pathology, Assiut University
Other Study IDs: 17300413
Record Dates: First submitted 2020-08-07; First posted 2020-08-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Coagulopathy
Keywords: hypercoagulable; COVID-19
MeSH Terms: conditions — Hemostatic Disorders; Thrombophilia; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Coagulopathy is one of the most significant prognostic factors in patients with COVID-19 and is associated with increased mortality and admission to critical care. Most commonly observed coagulopathy in patients hospitalized with COVID-19 (COVID-19-associated coagulopathy) is characterized by increased D-dimer and fibrinogen levels. 71% of patients who did not survive hospitalization reported to have developed disseminated intravascular coagulation (DIC) compared to 0.6% of survivors.

DETAILED DESCRIPTION:
studying the detailed coagulation screen and second line coagulation parameters including both thrombophilia screen and other acute phase coagulation factors.

ELIGIBILITY:
Inclusion Criteria:

* patients with COVID 19 positive by RT- PCR

Exclusion Criteria:

* no exclusions

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID 19 positive by RT- PCR who are admitted to Assiut University hospitals, Egypt.
  Age and sex matched controls
Sampling Method: Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Coagulation screen | 1 month
  Full coagulation screen
Thrombophilia screen | 1 month
  Full thrombophilia screen
VWF, FVIII | 1 month
  VWFAg, FVIII

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University Hospitals, Asyut, Egypt